CLINICAL TRIAL: NCT04298333
Title: Estimation of Maximum Tolerable Dose (MTD) and Minimum Efficient Dose (MED) of BP-C1 in Stage IV Breast Cancer Patients: A Phase I Dose-response Study
Brief Title: Dose-finding Study of BP-C1 in Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meabco A/S (Industry)
Collaborators: Meddoc (Other); Norwegian University of Life Sciences (Other); Meddoc Research Indonesia Ltd (Unknown); Meddoc Research Taiwan Ltd (Unknown)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: BMC2008-02
Record Dates: First submitted 2020-02-25; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Breast Cancer; Stage IV Breast Cancer
Keywords: BP-C1; Cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Benzene polycarboxylic acids complex with cis-diammineplatinum(II); Metastatic Breast Cancer; Platinum analogue; Metronomic chemotherapy; Breast cancer; Cisplatin; Cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will be open-label, multi-center with a sequential safety design based on 3-level between-patient Response Surface Pathway (RSP) algorithm. Three patients will be recruited consecutively to each sequence of three dose levels (dose level 1 - cumulative dose 0.64 mg/kg body weight, dose level 2 - cumulative dose 0.96 mg/kg body weight, dose level 3 - cumulative dose 1.12 mg/kg body weight).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BP-C1 (Experimental): BP-C1 will be used as supportive care
  Interventions: Drug: BP-C1

INTERVENTIONS:
Drug: BP-C1 — BP-C1, 0.05% solution for injection, will be administered intramuscularly once per day. The cumulative dose range will be 0.64-1.12 mg/kg body weight depending on design level (design level 1-3). The daily dose range will be 0.02-0.035 mg/kg body weight (0.04-0.07 mL/kg) depending on design level (design level 1-3).
  Dose level 1: 0.02 mg/kg body weight (0.04 mL/kg) intramuscularly once daily for 32 consecutive days; dose level 2: 0.03 mg/kg body weight (0.06 mL/kg) intramuscularly once daily for 32 consecutive days; dose level 3: 0.035 mg/kg body weight (0.07 mL/kg) intramuscularly once daily for 32 consecutive days.
  Changes in the cumulative dose of BP-C1 between patients in the sequence are predefined and will be adjusted by escalation/deescalation rules based on changes in toxicity observed in the previous design level.
  The duration of BP-C1 treatment will be 32 days.
  Other Names: Cis-coordinated complexes of platinum(II) with polymer of benzene polycarboxylic acids derived from lignin; Cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin

SUMMARY:
The purpose of this study is to estimate the cumulative Maximum Tolerated Dose (MTD) and Minimum Efficient Dose (MED) of BP-C1 in the short-term treatment of metastatic breast cancer patients.

DETAILED DESCRIPTION:
BP-C1, solution for injection 0.05%, is currently being developed for treatment of patients with metastatic breast cancer with palliative intent. Active substance of the product, which is a novel platinum-containing anticancer agent developed for intramuscular administration, is a cis-diammineplatinum(II) complexed with a polymer containing benzene polycarboxylic acids derived from lignin. The amphiphilic characteristics of the polymer have resulted in a product with clear and significantly altered and improved properties compared to other platinum analogues, e.g. cisplatin, carboplatin and oxaliplatin.

BP-C1 preserves antitumour activity of its predecessors (e.g. cisplatin and carboplatin), additionally offering the following advantages that ensure favourable outcome of treatment of metastatic breast cancer patients:

* injectable solution (intramuscular) does not cause injection site reactions;
* can be administered at home by a nurse or a patient;
* has an improved pharmacokinetic profile;
* demonstrates efficacy comparable to cisplatin and much higher than carboplatin (in-vitro; in-vivo data);
* exerts an additional immunomodulatory activity.

In this study BP-C1 will be administered as supportive care to patients with metastatic breast cancer (stage IV), who had undergone at least three lines of chemotherapy.

This study will be open-label, multi-centre with a sequential safety design based on 3-level between-patient Response Surface Pathway (RSP) algorithm. The eligible patients will be allocated to five independent sequences, with three patients in each sequence. The BP-C1 treatment period will be 32 days, the follow-up period will be 28 days after the last BP-C1 dose.

ELIGIBILITY:
Inclusion Criteria:

Female patients with histologically verified metastatic breast cancer (stage IV) with measurable metastases, between 18 and 80 years of age, who had undergone at least three lines of chemotherapy and had an expected survival time of at least 3 months.

Exclusion Criteria:

Patients fulfilling at least one of the following criteria will be excluded from participation in the study:

* Abnormal liver function classified as total bilirubin >34 μmol/L or ALAT > 3 times of the upper limit of normal (ULN). In case of metastases in the liver, the ALAT limit for exclusion is set to 5хULN.
* Abnormal kidney function defined by serum creatinine >120 μmol/L.
* Abnormal coagulation capacity defined by the relative arbitrary concentration of coagulation factors 2,7,10; INR >1.5.
* Verified metastases to the brain.
* Synchronous cancer except for non-melanoma skin cancer and early stage of cervical cancer.
* Abnormal haematology status defined by haemoglobin < 9.0 g/dL, platelet count < 100,000/mm^3 or leucocytes < 3x10^9/L.
* Clinically significant abnormal ECG.
* Karnofsky performance status score <60%.
* Pregnant or breast feeding women.
* Women of fertile age who do not want to be tested for possible pregnancy.
* Fertile female who do not want to use safe protection against pregnancy, starting one month before the start of the study treatment and lasting at least six weeks after.
* Uncontrolled bacterial, viral, fungal or parasite infection.
* Under systemic treatment with corticosteroids or other immunosuppressive drugs in the last 21 days before start of the trial treatment.
* Participating in another clinical trial with pharmaceuticals in the last six weeks before start of this trial treatment.
* Not able to understand information.
* Not willing or not able to give written consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06-27 (Actual); Primary Completion 2011-01-04 (Actual); Study Completion 2011-01-04 (Actual)

PRIMARY OUTCOMES:
Change in Maximum Common Terminology Criteria (CTC) score for Adverse Events | baseline to Day 32 of treatment and Day 28 of follow-up
  Maximum CTC score will be recorded using CTC v2.0 given as the highest observed CTC score at a given visit. The CTC scores will be recorded using CTC v2.0 divided in 15 System Organ Classes
Sum Common Terminology Criteria (CTC) score for Adverse Events | baseline to Day 32 of treatment and Day 28 of follow-up
  The Sum CTC score will be a sum of all registered CTC scores obtained at a given visit. The CTC scores will be recorded using CTC v2.0 divided in 15 System Organ Classes

SECONDARY OUTCOMES:
Number of registered Adverse Events (AEs) | baseline to Day 32 of treatment period and Day 28 of follow-up
Treatment Response | baseline to Day 32 of treatment and Day 28 of follow-up
  In accordance with RECIST v1.1 the treatment response will be classified as 'complete response', 'partial response', 'stable disease' or 'progressive disease': Complete response (CR): disappearance of all target lesions. Partial response (PR): at least 30% decrease in the sum of longest diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD): at least 20% increase in the sum of diameters of target lesions.
Proportion of patients with Disease Control Rate (DCR) | baseline to Day 32 of treatment and Day 28 of follow-up
  The DCR defined as patients classified as SD, PR, CR

CONTACTS AND LOCATIONS:
Locations (3):
- Sanglah University Hospital, Bali, Indonesia
- National Taiwan University Hospital, Taipei, Taiwan
- Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Benzene-Poly-Carboxylic Acids Complex with Cis-Diammineplatinum (II) Dichloride in the Treatment of Stage IV Breast Cancer Patients — http://benthamopen.com/ABSTRACT/TOBCANJ-5-7